CLINICAL TRIAL: NCT06906497
Title: A Phase IV, Non-randomized, Open-label Multinational Trial to Assess the Mechanism of Action for Lebrikizumab in Moderate-to-severe Atopic Dermatitis
Brief Title: Lebrikizumab in Moderate-to-severe Atopic Dermatitis
Acronym: ADfind
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johann E Gudjonsson MD PhD (Other)
Collaborators: Dermira, Inc. (Industry); Almirall, S.A. (Industry)
Responsible Party: Sponsor-Investigator, Johann E Gudjonsson MD PhD, Professor of Skin Molecular Immunology, Professor of Dermatology, Professor of Internal Medicine and Research Pr, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00261982
Record Dates: First submitted 2025-03-25; First posted 2025-04-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Moderate-to-severe Atopic Dermatitis (Experimental): A total of 48 subjects with active moderate-to-severe Atopic Dermatitis (AD) will be enrolled in a 60-week study from 4 independent sites (2 US sites and 2 EU sites).
  Interventions: Drug: lebrikizumab

INTERVENTIONS:
Drug: lebrikizumab — Patients will receive lebrikizumab with a 500 mg loading dose administered subcutaneously at baseline and Week 2 followed by 250 mg every 2 weeks until Week 24.
  At week 24, patients with ≥ Eczema Area and Severity Index (EASI) 50 will continue in the study and begin receiving lebrikizumab 250mg every 4 weeks (Q4W), while patients with <EASI 50 will be discontinued from the study.
  At week 36, patients with EASI ≥50 to <90 will remain on Q4W through W60 (do not enter withdrawal arm), while patients with sustained low disease activity (IGA 0/1 or EASI≥90 response for at least 3 months assessed at W24 and W36) will withdraw from lebrikizumab treatment
  Other Names: Ebglyss

SUMMARY:
This research is studying a drug already approved for the treatment of atopic dermatitis (AD). This research collects health-related information and blood and skin samples to understand if the study drug, lebrikizumab, leads to long-term improvement in AD skin.

DETAILED DESCRIPTION:
Lebrikizumab, the drug used in the study, has been deemed IND exempt by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of AD for at least 1 year before the screening visit and topical treatment was inadequate or inadvisable.
* Moderate-to-severe AD with involvement > 10% of body-surface-area (BSA) and investigator global assessment (IGA) score =3 (based on the IGA scale ranging from 0 to 4, in which 3 is moderate and 4 is severe) at both the screening and baseline visits.
* Subject has an Eczema Area and Severity Index (EASI) score =16 at screening and baseline.
* Subject has a pruritus NRS =4.
* Subject is biologic naïve.
* Female subjects of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree either to commit to true abstinence throughout the study and for at least 17 weeks after the last study drug (SD) injection, when this is in line with the preferred and usual lifestyle of the subject, or to use a highly-effective and approved method of contraception throughout the study and for at least 17 weeks after the last study drug injection.
* Subject willing and able to comply with all of the clinical study protocol's time commitments and procedural requirements.
* Understand and sign an informed consent form (ICF) (and assent form, when applicable) before any investigational procedure(s) are performed.

Exclusion Criteria:

* Previous treatment with lebrikizumab or participation in a lebrikizumab study.
* History of anaphylaxis as defined by the Sampson criteria.
* Treatment with topical corticosteroids, calcineurin inhibitors, Jak inhibitors, or crisaborole within 1 week prior to the baseline visit.
* Prior treatment with dupilumab or tralokinumab.
* Treatment with any of the following agents within 4 weeks prior to the baseline visit:

  1. Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-., Janus kinase inhibitors (JAKi), azathioprine, methotrexate).
  2. Phototherapy and photochemotherapy (PUVA) for AD.
* Treatment with the following prior to the baseline visit:

  1. An investigational drug within 8 weeks or 5 half-lives (if known), whichever is longer.
  2. Cell-depleting biologics, including to rituximab, within 6 months.
  3. Other biologics within 5 half-lives (if known) or 16 weeks, whichever is longer.
* Use of prescription moisturizers within 7 days of the baseline visit.
* Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit.
* Treatment with a live (attenuated) vaccine within 12 weeks of the baseline visit or planned during the study.
* Uncontrolled chronic disease that might require bursts of oral corticosteroids, e.g., co-morbid severe uncontrolled asthma requiring systemic [oral and/or parenteral] corticosteroid treatment or hospitalization for > 24 hours).
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, anti-parasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit. NOTE: patients may be rescreened after infection resolves.
* Evidence of active acute or chronic hepatitis (as defined by the Department of Health & Human Services Centers for Disease Control and Prevention) or known liver cirrhosis.
* Diagnosed active endoparasitic infections or at high risk of these infections.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per the Investigator's judgment.
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* In the Investigator's opinion, any clinically significant laboratory results from the chemistry, hematology or urinalysis tests available in the medical history.
* Presence of skin comorbidities that may interfere with study assessments.
* History of malignancy, including mycosis fungoides, within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
* Severe concomitant illness(es) that in the Investigator's judgment would adversely affect the patient's participation in the study. Any other medical or psychological condition that in the opinion of the Investigator may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient because of his/her participation in this clinical trial, may make patient's participation unreliable, or may interfere with study assessments.

  20. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Degree of normalization of transcriptomic/epigenetic profile | Up to week 60
  Assessed from skin biopsies using the molecular response to lebrikizumab among patients with atopic dermatitis

SECONDARY OUTCOMES:
Molecular response to Lebrikizumab | weeks 36 to 60
  Assessed from skin biopsies using the molecular response to lebrikizumab among patients with atopic dermatitis, analyzed for those who discontinued treatment as well as those who continued it
Skin barrier function | Up to week 60
  Assessed by serial transepidermal water loss (TEWL) measurements in lesional skin. TEWL will be measured using Courage + Khazaka gmbh tewameter hex for spot measurements
Clinical response as assessed be the Eczema Area and Severity Index (EASI) | Up to week 60
  Clinical response assessed using the EASI - Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicating greater severity of AD to be correlated with Molecular response, assessed using single-cell RNA-sequencing
  This will be done using correlation based analyses and with correction for multiple testing (FDR).
Clinical response as assessed using the investigator global assessment (IGA) | Up to week 60
  Clinical response assessed using the IGA - Score ranges from '0' = Clear to '5' = Very Severe Disease to be correlated with molecular response, assessed using single-cell RNA-sequencing.
  This will be done using correlation based analyses and with correction for multiple testing (FDR).
Clinical response as assessed using the Peak Pruritus Numerical Rating Scale (NRS) (Pruitis NRS) | Up to week 60
  Clinical response assessed using the Pruitis NRS - is a single self-report item on an 11-point scale (0 to10) where 0 is No itch, and 10 is the Worst itch imaginable. That will be correlated with the molecular response, assessed using single-cell RNA-sequencing
  This will be done using correlation based analyses and with correction for multiple testing (FDR).

CONTACTS AND LOCATIONS:
Overall Officials: Johann E. Gudjonsson, MD, PhD, Principal Investigator — University of Michigan
Locations (4):
- United States (2):
  - Physioseq USA - CA, Folsom, California
  - University of Michigan, Ann Arbor, Michigan
- University of Freiburg, Freiburg im Breisgau, Germany
- Lausanne University Hospital, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No